CLINICAL TRIAL: NCT02337296
Title: An Intervention to Promote Oral Agent Adherence and Symptom Management: ADHERE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Huron Medical Center (Other); Allegiance Health (Other); Sparrow Health System (Other)
Responsible Party: Principal Investigator, Sandra Spoelstra, Assistant Professor, Michigan State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC103421
Record Dates: First submitted 2014-11-20; First posted 2015-01-13 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Cancer
Keywords: Motivational Interviewing; Cognitive Behavioral Therapy; Cancer; Oral Agents; Adherence
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1 - Intervention (Other): Five patients will be enrolled consecutively for the ADHERE intervention and be followed in order to refine the intervention as needed. This permits the investigation of the process of change at baseline, after the intervention, and across the phases.
  Interventions: Behavioral: ADHERE
- Phase 2 - Control Group (No Intervention): Following completion of Phase 1 and prior to initiation of enrollment in the intervention group, patients will be enrolled in the control group and will receive usual care.
- Phase 2 - Intervention Group (Experimental): Following enrollment of all control group patients, the intervention group will be recruited and enrolled and the ADHERE intervention will be conducted by the trained APRN interventionist at cancer center.
  Interventions: Behavioral: ADHERE

INTERVENTIONS:
Behavioral: ADHERE — ADHERE entails a face-to-face 30 minute session during week 1 while in the clinic/office and three subsequent ADHERE phone calls for 10 minutes each, weekly during weeks 2-4 to promote symptom management and adherence to their oral agent regimen. The face-to-face intervention and phone interactions will consist of Motivational Interviewing and Cognitive Behavioral Therapy interaction strategies. Each patient will be given a Medication Management and Symptoms Management Toolkit, to assist with symptom management at home.
  All patients (intervention and control) receive weekly assessments of symptom severity and oral agent adherence (weeks 2-7). At exit (week 8), all patients receive an assessment of depressive symptoms, self-efficacy, beliefs, motivation, symptom severity, and adherence.
  Arms: Phase 1 - Intervention; Phase 2 - Intervention Group

SUMMARY:
This study includes a novel intervention entitled "ADHERE," which includes one semi-structured 30-minute face-to-face session and three 10-minute weekly phone sessions over 4 weeks, administered by an advanced practice nurse (APRN) to promote management of symptoms and adherence in patients prescribed oral anti-cancer agents. Innovations in cancer treatment are changing the treatment delivery landscape. It is projected that by 2015, 25% of treatment will be delivered in pill form. This shift in the treatment paradigm places greater responsibility on patients. However, patients with cancer are known to miss as much as one-third of the prescribed doses of oral agents required for treatment of their disease. Barriers to oral agent adherence include symptom severity, low self-efficacy, depressive symptoms, lack of motivation, or beliefs that the medicine will not help, age, and regimen complexity. The therapeutic outcome for those taking oral agents depends heavily on the ability of patients to adhere to the prescribed regimen. Thus, a critical need exists to test interventions that promote adherence and symptom management in patients taking oral agents.

ADHERE provides systematic patient education (PE) with the investigators evidence-based Medication Management and Symptom Management Toolkit (Toolkit). This is combined with brief cognitive behavioral therapy (CBT) to focus thoughts and beliefs to influence action; and motivational interviewing (MI) to elicit reasons from patients to take action. The National Cancer Institute (NCI), American Society of Clinical Oncology (ASCO), and Oncology Nursing Society (ONS) have made adherence to oral agents a priority. Thus, the investigators are testing ADHERE's impact on symptom severity and adherence to the oral agent regimen and determining the acceptability and feasibility of the intervention among patients with cancer.

DETAILED DESCRIPTION:
Purpose/Aims: Over 50 oral agents in pill form are currently on the market, with projections that in three years, 25% of cancer treatment will be delivered in pill form with patients assuming responsibility for self-management at home. For oral agents to achieve a therapeutically effective level for cancer treatment, patients must strictly adhere to the regimen. Adherence to oral cancer agents is often less than 80%, which may be inadequate for treating the cancer. The aim of this study is to refine and determine the feasibility and preliminary efficacy of an intervention (entitled "ADHERE") that uses motivational interviewing (MI) to elicit reasons to adhere and brief cognitive behavioral therapy (CBT) as a mechanism for goal-oriented systematic patient education (PE) to promote adherence and symptom management among cancer patients prescribed oral agents. Significance: This study targets a challenging clinical problem among patients with a life-threatening disease, assisting them in adhering to and completing their cancer treatment, impacting symptoms, quality of life, and longevity. Framework: The Motivation and Behavior Skills Model guides this work. The model asserts even a well informed or highly motivated patient will have difficulty achieving and sustaining optimal adherence if they lack the skills required to acquire or self-manage or feel incapable of performing such behaviors. Main Variables: Adherence and symptom severity. Methods: This practice-based study will be conducted using a 4-week intervention (ADHERE) to promote adherence and symptom management in patients newly prescribed oral agents in two phases. Phase 1 will use a single-subject-design to consecutively enrolling 5-patients from a cancer center over 4-weeks and investigators will use an iterative process to refine ADHERE in a practice-based setting. Phase 2 will use an 8-week quasi-experimental sequential design, enrolling 60-patients (30 intervention & 30 control) from 2-cancer centers to examine feasibility and preliminary efficacy of a 4-week ADHERE intervention and follow-up for 4-weeks to assess adherence and symptom management. Descriptive statistics will be provided as appropriate for all data collected, and 95% confidence intervals will be provided by using exact method for outcome variables, such as: the proportion of patients who are enrolled to participate in the study among those who are recruited; the proportion of ADHERE received by the patient over the four-week time period; and the proportion of patients who report high satisfaction with ADHERE. Exploratory analysis of efficacy as measured weekly by proportion of pills taken compared to what was prescribed. Implications: This study has the potential to have a transformative impact on oral agent adherence by developing an advanced practice registered nurse-led strategy to promote adherence among the increasing number of cancer patients who receive their cancer treatment in pill form. This intervention will lead to standardized care for patients newly prescribed oral agents. Results of this study will be used to inform the development of an R01 application to conduct a larger randomized trial to test the efficacy of this innovative intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer
* Newly prescribed (within 60-days) an oral anti-cancer agent
* Have a phone and be willing and able to receive phone calls
* Able to read, speak, and understand English
* Cognitively intact and able to self-manage and follow direction, as evaluated by the Recruiter

Exclusion Criteria:

* Unable to accept phone calls

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Proof-of-concept of the ADHERE intervention among patients who are on oral agents. | Calculated at the end of study (at 8-weeks)
  Indices used to evaluate proof-of-concept include proportion of those enrolled among all recruited, the proportion of those who complete the intervention among all enrolled into the intervention group, and proportion of those satisfied among those who complete the intervention.

SECONDARY OUTCOMES:
Preliminary efficacy of the ADHERE intervention on adherence to oral agents. (proportion of pills taken compared to what was prescribed and will be considered continuous variables) | Calculated at the end of study (at 8-weeks)
  The primary efficacy outcome of the intervention will be oral agent adherence as measured weekly by proportion of pills taken compared to what was prescribed and will be considered continuous variables. Total proportion of pills taken will also be calculated as a measure, i.e., the total number of pills taken divided by total number of pills prescribed.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra L Spoelstra, PhD, RN, Principal Investigator — Michigan State University
Locations (2):
- United States (2):
  - Allegiance Health, Jackson, Michigan
  - Huron Medical Center, Port Huron, Michigan